CLINICAL TRIAL: NCT04916262
Title: Correlation Between TCM Syndrome Factors and TSH Changes of Thyroid Hormone Withdrawal Before Iodine Therapy in Postoperative Patients With Thyroid Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: LJB-02
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Differentiated Thyroid Carcinoma; TCM Syndrome Type
Keywords: Differentiated Thyroid Carcinoma; TCM syndrome type

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TSH < 30uIU/mL group: Clinical information was collected from patients with TSH < 30UIU /mL on the 14th day of thyroxine withdrawal before 131I treatment，including TCM syndrome elements, general information ,medical history and biochemical examination during hospitalization.
- TSH ≥ 30uIU/mL group: Clinical information was collected from patients with TSH ≥ 30UIU /mL on the 14th day of thyroxine withdrawal before 131I treatment，including TCM syndrome elements, general information ,medical history and biochemical examination during hospitalization.

SUMMARY:
The purpose of this study is to make a dialectical classification of patients who will receive 131I treatment after operation of thyroid cancer from the point of view of dialectics of syndrome elements of traditional Chinese medicine. By observing the changes of TSH among patients with different syndrome types, investigators can better understand the reasons for the differences in TSH changes among patients. Thus, it provides a basis for putting forward the scheme of stopping taking levothyroxine before iodine treatment, improving the quality of life of patients after radical thyroidectomy, and providing reference for individualized guidance of the timing of radioactive iodine therapy for patients after DTC.

DETAILED DESCRIPTION:
Thyroid cancer is a common thyroid tumor. In the past few decades, the incidence of thyroid cancer in most parts of the world has increased steadily year by year. At present, the best treatment for differentiated thyroid cancer at home and abroad is surgery + radioactive iodine + thyroid hormone replacement inhibition.131I therapy, as an important adjuvant therapy for patients with DTC, can effectively remove the residual thyroid tissue and unresectable local and distant metastatic lesions during the operation.

It is considered that the level of TSH and the time of thyroid hormone withdrawal are important factors affecting the efficacy of radioiodine therapy, and there is a close relationship between the two factors. Clinically, investigators also observed that TSH changes were different in patients who were about to receive iodine treatment after DTC during the withdrawal of thyroxine. In some patients, TSH levels rise rapidly in a short period of time, while others rise slowly. For patients with rapid increase of TSH (sometimes even more than 100uIU/ml), it may promote tumor growth, recurrence and recessive metastasis. Patients with slow rise of TSH may need to constantly review thyroid function until reaching the standard, which brings inconvenience to patients, and withdrawal of drugs for too long will affect patients' physical, psychological and living conditions, resulting in patient discomfort.

In this study, the dialectical classification of TCM syndrome factors was carried out in the patients before radioiodine therapy after DTC. After collecting the patients who met the inclusion and exclusion criteria, they were divided into two groups according to TSH ≤ 30uIU/mL and TSH > 30uIU/mL on the 14th day. The TCM syndrome elements and other clinical information of each group were collected respectively. Investigators will observe the changes of TSH in patients with different types of TCM syndrome factors, and gain a deeper understanding of the reasons for the differences in TSH changes. Investigators hope to provide a basis for putting forward a plan to stop thyroxine before iodine therapy, to improve the quality of life of postoperative patients with thyroid cancer, and to provide a reference for individualized guidance of the timing of radioactive iodine therapy for patients after DTC.

ELIGIBILITY:
Inclusion Criteria:

1. Study time: June 1, 2021, to January 1, 2022;
2. Study site: The First Affiliated Hospital of Shandong First Medical University;
3. 18-75 years old (including upper and lower limits), male or female;
4. Patients with differentiated thyroid carcinoma diagnosed pathologically after total thyroidectomy
5. Patients with oral levothyroxine tablets ≥ 4 weeks after operation
6. Patients who have stopped taking levothyroxine tablets and whose TSH < 4.2uIU/ml at the time of withdrawal
7. Patients who meet the 131I treatment criteria

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with various mental disorders, unconscious, etc.
3. Cases with inaccurate information collection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid cancer who need 131I therapy after operation
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure 1 | The data will be collected, analyzed and calculated in about 3 days.
  The TCM syndrome types of patients participating in this study were evaluated by TCM syndrome factor scale, and the diagnosis was established when the total weight of the scale was more than 20
Primary Outcome Measure 2 | The data will be collected, analyzed and calculated in about 3 days.
  Correlation analysis was used to analyze the correlation between TCM syndrome types and the time needed for thyrotropin ≥ 30uIU/ml during the treatment of thyroid hormone withdrawal.

SECONDARY OUTCOMES:
Secondary Outcome Measure 1 | 2 weeks.
  To observe the TSH≥30uIU/mL rate after Withdrawal of Suppressive Thyroxine Therapy 2 weeks in Preparation for Radioactive Iodine Administration to Patients with differentiated thyroid cancer.
Secondary Outcome Measure 2 | 2 weeks.
  Correlation analysis was used to analyze the effect of age (in years) on the level of serum TSH after thyroxine withdrawal treatment.
Secondary Outcome Measure 3 | 2 weeks.
  The effect of gender on serum TSH level after thyroxine withdrawal treatment was analyzed by correlation analysis.
Secondary Outcome Measure 4 | 2 weeks.
  Height and weight measurement instrument (HW-900Y) was used to measure height (in meters). Correlation analysis was used to analyze the effect of height on serum TSH level after thyroxine withdrawal treatment.
Secondary Outcome Measure 5 | 2 weeks.
  The height and weight meter (HW-900Y) was used to measure the body weight (in kilograms), and the correlation analysis was used to analyze the effect of weight on the level of serum TSH after thyroxine withdrawal treatment.
Secondary Outcome Measure 6 | 2 weeks.
  weight and height will be combined to report BMI in kg/m^2.Correlation analysis was used to analyze the effect of BMI on serum TSH level after thyroxine withdrawal therapy.
Secondary Outcome Measure 7 | 2 weeks.
  Total cholesterol detection kit (COD-PAP) was used to measure serum cholesterol (in mmol/l). Correlation analysis was used to analyze the effect of serum cholesterol on serum TSH level after thyroxine withdrawal treatment.
Secondary Outcome Measure 8 | 2 weeks.
  Serum triglyceride (mmol/l) was detected by triglyceride determination kit (GPO-PAP). The effect of serum triglyceride on serum TSH level after thyroxine withdrawal treatment was analyzed by SPSSstatistics20.0.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Liao, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital

REFERENCES:
- [Background] Zhou Y, Yang Y, Zhou T, Li B, Wang Z. Adiponectin and Thyroid Cancer: Insight into the Association between Adiponectin and Obesity. Aging Dis. 2021 Apr 1;12(2):597-613. doi: 10.14336/AD.2020.0919. eCollection 2021 Apr. PMID 33815885
- [Background] Stewart LA, Kuo JH. Advancements in the treatment of differentiated thyroid cancer. Ther Adv Endocrinol Metab. 2021 Mar 17;12:20420188211000251. doi: 10.1177/20420188211000251. eCollection 2021. PMID 33796254
- [Background] Borges de Souza P, McCabe CJ. Radioiodine treatment: an historical and future perspective. Endocr Relat Cancer. 2021 Sep 3;28(10):T121-T124. doi: 10.1530/ERC-21-0037. No abstract available. PMID 33690155
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967